CLINICAL TRIAL: NCT06349213
Title: Uncovering the Cognitive and Neural Mechanisms Underlying Cognitive Time
Acronym: TIMES
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C23-19; 2023-A02263-42 (Other: Secondary ID)
Record Dates: First submitted 2024-03-21; First posted 2024-04-05 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Young healthy volunteers: Healthy young adults (20-35 years) will undergo the first two visits detailed above.
  Interventions: Radiation: FDOPA injection before PET imaging; Behavioral: Time perception tasks; Device: fMRI imaging; Device: EEG imaging
- Older healthy volunteers: Healthy older adults (60-85 years) will undergo each visit detailed above (five visits in total).
  Interventions: Radiation: FDOPA injection before PET imaging; Behavioral: Time perception tasks; Device: fMRI imaging; Device: EEG imaging; Behavioral: 3 year follow-up

INTERVENTIONS:
Radiation: FDOPA injection before PET imaging — Fluorodopa labelled with fluorine 18 (physical half-life of 109.6 min) is used at a dosage of 1 to 2 MBq/kg in neuroimaging, depending on the sensitivity of the PET camera used. For these reasons, a dose of 2 MBq/kg will be administered slowly intravenously (approximately 1 minute for a maximum bolus of 10 mL). PET acquisitions will be performed at 90 minutes post-injection and will last 30 minutes. Participants will be asked to have fasted for at least 4 hours at the time of injection, with no restriction on fluid intake.
Behavioral: Time perception tasks — The main tasks involves the comparison of duration to assess aging effects on the precision of temporal representations
Device: fMRI imaging — Imaging of brain structure during the completion of the time perception task
Device: EEG imaging — Recording of neural dynamics during the completion of the time perception task
Behavioral: 3 year follow-up — Behavioral and EEG follow-up (for older adults only)
  Groups: Older healthy volunteers

SUMMARY:
Time processing, the ability to process and encode temporal information, is essential for cognitive functioning and for a large number of daily life activities. In particular, the processing of durations of several seconds is central to cognition, impaired in several pathologies, and has been associated with cognitive changes with advancing age. While behavioral studies have been conducted to specify the neural bases of temporal cognition and their association with other cognitive functions, the mechanisms underlying age-related changes, and individual differences, remain unknown. The project will characterize ageing effects on timing mechanisms and their neural underpinnings. Building on recent advances from neuroscience and age-related cognitive changes, the project focuses on the precision of duration processing, that declines with age, and the associated neural bases. Participants will perform a duration judgement task while (a) electroencephalography, and (b) functional magnetic resonance imaging activity are simultaneously recorded to investigate age effects on structural and functional network connectivity. In addition, striatal dopamine will be measured using a FDOPA PETscan. Evaluation of other temporal cognition processes and general cognition will also be performed. This combination offers a unique opportunity to accurately specifying the neurophysiological underpinning of aging effects on time processing changes. This project will further our understanding of the variability of cognitive performance with advancing age, and contribute to identifying new measures of temporal impairments.

DETAILED DESCRIPTION:
The main research examinations for all participants will be divided into two initial visits (V1: approximately 3.5 hours and V2: approximately 2.5 hours) at the GIP Cyceron (neuroimaging center) premises.

As part of the longitudinal follow-up, older participants only will complete one follow-up session (visits: V3, V4 and V5) of approximately two and a half hours per year at the PMRCI premises, for three years after visit 2.

During the various visits, participants may be accompanied by a support person of their choice.

The first visit will last approximately 3 and a half hours and will consist of two parts:

- First part of visit 1: Inclusion medical visit (V1, GIP Cyceron) The first part of Visit 1 will be carried out at GIP Cyceron after a cooling-off period of at least 7 days from the day of the telephone interview and will last approximately 1 hour. It will begin with the information and consent procedure carried out by an investigator registered with the Order of Physicians or his or her designated representative and registered on the task delegation list. Participants will be informed of the purpose, recipients and retention periods for all data collected as part of their participation in the research.

Prior to signing the consent form, the eligibility criteria (inclusion and non-inclusion criteria) will be checked by the investigator. The visit also includes the taking of a medical history and current treatments.

- Second part of Visit 1 (V1, GIP Cyceron): simultaneous EEG-fMRI, neuropsychological assessment : The second part of the V1 visit will be carried out at GIP Cyceron and will last approximately 2 and a half hours. It will begin with a urine pregnancy test for women of childbearing age and verification that there are no contraindications to the MRI examination. The EEG-MRI imaging will then last approximately 1.5 hours, followed by a 15-30 minute break. Finally, the neuropsychological evaluation will last about an hour and will include the performance of some of the neuropsychological tests and self-questionnaires in the presence of members of the investigating team. The tests and self-questionnaires will last approximately one hour and will be adjusted according to each individual's completion time and any level of fatigue.

During this visit, participants will perform a temporal judgement task while EEG and fMRI functional data are being recorded. Anatomical data will also be collected. The accuracy of time processing will be assessed in the MRI using bisection and temporal generalisation tasks.

Visit 2 (V2, GIP Cyceron, maximum one month after V1): PET scan and neuropsychological assessment The V2 visit will be carried out at GIP Cyceron approximately one month after visit 1 and will last about 2 and a half hours. A telephone call from the project leader will enable this visit to be scheduled. Participants will be asked to have fasted for at least 4 hours at the time of the visit, with no restriction on fluid intake. The visit will begin with PET imaging for approximately 1.5 hours, followed by a 15-30 minute break. For women of childbearing age, a urine pregnancy test will be performed prior to the PET scan. The neuropsychological assessment described in V1 will also be carried out for approximately one hour, in the presence of members of the investigating team.

The dopaminergic status of the nigrostriatal pathway will be explored in vivo using a Discovery RX VCT 64 whole-body PET-CT scanner (General Electric Healthcare; maximum axial FAV 50cm). The investigator will use [18F]-FDOPA (DOPACIS®), a fluorine-18 labelled radiopharmaceutical. This radiopharmaceutical indirectly reflects the number of dopaminergic neurons via the enzymatic activity of dopa-decarboxylase within these neurons.

Visits 3, 4, 5 (PMRCI, approximately once a year following V2):

The procedure for these three visits is identical. Participants will be contacted by the project leader to plan these visits. Only elderly participants will be included in the longitudinal follow-up. The elderly participants will first perform the temporal judgement task performed in V1 while the EEG activity is being recorded (approximately 1.5 hours). Following a 15-30 minute break, all the neuropsychological measures (tests and self-questionnaires) described above will be carried out (approximately 1.5 hours). These visits will take place one, two and three years after the second visit. Only older individuals will be included in the longitudinal follow-up in order to identify the factors associated with the variability of cognitive trajectories, which is greater during the ageing process.

At each follow-up visit (visits 3, 4 & 5), the investigator will check that the participant is not under legal protection (guardianship, curators or safeguard of justice) as well as the absence of global cognitive deficit attested by a score on the MOCA scale greater than or equal to 26/30. If this is the case, the participant will not be able to continue to take part in the research. The tutor/supervisor will be informed of this condition.

ELIGIBILITY:
Inclusion Criteria:

1. Membership of a social security scheme or beneficiary of such a scheme.
2. At least 7 years' schooling.
3. Acceptance and signature of the informed consent form
4. Fluency in French (as assessed by the project leader)
5. Age between 20 and 35 years inclusive for young healthy subjects, and between 60 and 85 years inclusive for elderly healthy subjects.
6. Effective contraception for women of childbearing age: Contraception will be considered effective from the moment the participant declares taking an oral contraceptive, the presence of an IUD, diaphragm or contraceptive implant, or the performance of a tubal ligation or sterilisation.
7. Absence of global cognitive deficit attested by a score on the MOCA scale greater than or equal to 26/30.

Exclusion Criteria:

1. Persons under guardianship, curators or safeguard of justice.
2. Pregnant women, women in labor and nursing mothers
3. Chronic neurological conditions
4. Uncorrected visual difficulties
5. Encephalitis
6. Endocrine or liver disease
7. History of head trauma with loss of consciousness lasting more than one hour
8. History of cancer in the last 5 years, with the exception of squamous cell carcinoma of the skin
9. Presence or history of chronic alcoholism or drug addiction
10. Presence of clinically significant major psychiatric disorders (according to DSM-IV-TR criteria) or symptoms that could affect the participant's ability to complete the research.
11. Use of medications that may modulate the dopaminergic system (psychotropic, with the exception of sleeping pills or occasional use of anxiolytics, as decided by the principal investigator).
12. Contraindications to MRI examination (pregnancy; pacemaker or neurosensory stimulator or implantable defibrillator; clip on an aneurysm or clip on a vascular malformation of the brain; intraocular or cerebral ferromagnetic foreign body; prosthesis or mobilizable ferromagnetic metal object or splinter; cochlear implant ; peripheral stimulator; neurosurgical ventriculoperitoneal shunt valves; permanent eyelid or lip make-up; jewelry or piercing that cannot be removed; certain tattoos depending on the type of ink, size and location; automated injection devices such as insulin pumps, blood glucose sensors, claustrophobia).
13. Radiotracer contraindications: Hypersensitivity to product excipients, chronic alcoholism, kidney disease.
14. Participation in research involving exposure to ionizing radiation (nuclear medicine or radiology examinations) in the year preceding inclusion or during a period of exclusion from other research.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participant with no diagnosed condition
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
EEG phase lag index differences between group | Through study completion, an average of 3 years
  Functional connectivity (EEG phase lag index (PLI) in each frequency band) differences between young and older adults during completion of the duration comparison task

CONTACTS AND LOCATIONS:
Locations (1):
- Cyceron Boulevard Henri Becquerel, Caen, France

IPD SHARING:
Plan to Share IPD: No